CLINICAL TRIAL: NCT00978653
Title: Prospective Study of Allopurinol Treatment That Improves Endothelial Function by Decreasing Uric Acid Levels of Patients With Chronic Kidney Disease
Brief Title: The Effect of Uric Acid Decrement on Endothelial Function in Patients With Chronic Renal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Alaattin Yildiz, Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 200931386
Record Dates: First submitted 2009-09-14; First posted 2009-09-17 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Hyperuricemia; Chronic Kidney Disease
Keywords: allopurinol; chronic kidney disease; endothelial dysfunction; hyperuricemia; uric acid; vascular endothelium; xanthine oxidase inhibitor
MeSH Terms: conditions — Hyperuricemia; Renal Insufficiency, Chronic | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allopurinol (Experimental): Hyperuricemic (uric acid (UA)>7 mg/dL), nondiabetic CKD patients without any comorbidity, age<60 years with creatinine clearance (CrCl) between 20 and 60ml/min were evaluated.
  Interventions: Drug: allopurinol

INTERVENTIONS:
Drug: allopurinol — 150 mg once a day
  Other Names: urikoliz

SUMMARY:
In this prospective study, the investigators aimed to evaluate the effects of improved hyperuricemia, a minor cardiovascular risk factor, on endothelial dysfunction in patients with chronic kidney disease.

DETAILED DESCRIPTION:
Endothelial dysfunction (ED) is a key event in the development of atherosclerotic cardiovascular disease observed in patients with chronic kidney disease (CKD). Experimental models have shown that hyperuricemia causes hypertension and renin angiotensin system activation. In this prospective study, the investigators aimed to evaluate the effects of improved hyperuricemia, a minor cardiovascular risk factor, on ED in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory finding of hyperuricemia
* Patients between ages of 18 and 60 years
* Non-diabetic patients
* Creatinine clearance values between 20 and 60 mL/min/1.73 m2

Exclusion Criteria:

* Low (< 20 ml/min/1.73 m2) creatinine clearance,
* Patients with diabetes mellitus, ischemic heart disease, acute coronary syndrome, congestive heart failure (CHF) (New York Heart Association class II or greater), valvular heart disease and a history of cerebral infarction or transient ischemic attack.
* Patients taking urate lowering medication (allopurinol and probenecid)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Endothelial function improvement with uric acid lowering treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Berna Yelken, MD, Principal Investigator — Division of Nephrology, Istanbul Faculty of Medicine, Istanbul University; Yasar Caliskan, Principal Investigator — Division of Nephrology, Istanbul Faculty of Medicine, Istanbul University; Alaattin Yildiz, Prof, MD, Study Director — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul University; Numan Gorgulu, MD, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul University
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)